CLINICAL TRIAL: NCT02574403
Title: Multicentric, Prospective Open-label Study Assessing an Algorithm-based Strategy of Eculizumab Discontinuation in Children and Adults With Atypical Hemolytic Uremic Syndrome (aHUS)
Brief Title: Study Assessing an Algorithm-based Strategy of Eculizumab Discontinuation in Children and Adults With aHUS
Acronym: STOPECU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC15_0061
Record Dates: First submitted 2015-10-05; First posted 2015-10-12 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Atypical Hemolytic Uremic Syndrome
Keywords: atypical hemolytic uremic syndrome (aHUS); eculizumab discontinuation
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- without eculizumab (Experimental)
  Interventions: Drug: eculizumab

INTERVENTIONS:
Drug: eculizumab — eculizumab discontinuation

SUMMARY:
Atypical hemolytic syndrome (aHUS) is a severe renal disease affecting children and adults. It is characterized by the occlusion of intrarenal vessels due to the presence of platelet/fibrin thrombi, and leads to end-stage renal disease in up to 2/3 of patients. The discovery of complement alternative pathway as a major risk factor for aHUS has led to the design of a disease-specific treatment, the anti-C5 monoclonal antibody, eculizumab. Complement inhibition using eculizumab has clearly improved the renal outcome of aHUS patients with a dramatic decrease in the risk of end-stage renal disease. However, the optimal duration of eculizumab therapy is still debated. The present study aims to assess the feasibility and safety of the discontinuation of eculizumab treatment in children and adults with aHUS.

DETAILED DESCRIPTION:
A visit (physical examination; blood pressure measurement) will be performed every month for 3 months, and every 3 months for 21 months.

Blood (serum creatinine, platelet count, hemoglobin, LDH, haptoglobin) and urine (proteinuria/creatininuria ratio and microscopic hematuria) tests will be performed every 2 weeks from inclusion to M6 and subsequently every month starting M7 Urine dipstick (for albuminuria and microscopic hematuria) will be performed by the patients at home at least twice a week.

Markers of complement activation and biomarkers of endothelial cells activation and immune cells activation will be assessed at baseline, M1, M3, M6, M9, M12, M18 and M24.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adults under eculizumab treatment for aHUS (initial episode or relapse) defined by at least two of the following: thrombocytopenia (platelet count < 150 G/L), mechanical hemolytical anaemia (Hb < 10 g:dl, LDH > upper limit of normal, undetectable haptoglobin, presence of schizocytes on blood smear), acute kidney injury (serum creatinine and/or proteinuria/creatininuria > upper limit of normal for age or an increase > 15% compared to baseline levels )
2. Patients not requiring dialysis.
3. Adults: HUS remission and normal or stabilized renal function under eculizumab treatment since at least 6 months (3 months in patients with MCP mutations)
4. Children: age > 3 years at eculizumab withdrawal; HUS remission and normal renal function under eculizumab treatment since at least 3 months in children with isolated MCP mutation, at least 6 months in children with complement mutation other than MCP.

Exclusion Criteria:

1. Patients on dialysis.
2. Women treated with eculizumab starting or planning a pregnancy. Pregnancy including the post-partum period is high-risk periods for the occurrence of aHUS.
3. Patients who did not give informed consent.
4. Patients under protection of a judicial authority

Patients can be enrolled in the study within ten weeks after Eculizumab stop.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
The incidence of aHUS relapse during 2 years of follow-up after eculizumab discontinuation | 24 months
  aHUS relapse will be defined by the coexistence of at least two of the following:
  * thrombocytopenia (platelet count < 150 G/L),
  * mechanical hemolytical anaemia (Hb < 10 g/dl, LDH > upper limit of normal, undetectable haptoglobin, presence of schizocytes on blood smear),
  * acute kidney injury (serum creatinine and/or proteinuria/creatininuria > upper limit of normal for age or an increase > 15% compared to baseline levels ),
  * features of thrombotic microangiopathy (glomerular and/or arteriolar thrombi, doubles contours, endothelial cells detachment) in a kidney biopsy, if performed.

CONTACTS AND LOCATIONS:
Overall Officials: Fadi FAKHOURI, Pr, Study Director — Nantes CHU
Locations (22):
- France (22):
  - CHU Amiens, Amiens
  - CHU Bordeaux, Bordeaux
  - CHU Caen, Caen
  - CH métropole Savoie, Chambéry
  - CH Dijon, Dijon
  - Ch Le Mans, Le Mans
  - CHRU Lille, Lille
  - CHU lyon, Lyon
  - AP-HM, Marseille
  - CH Metz Thionville, Metz
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - BICHAT, Paris
  - Hopital Necker, Paris
  - Hopital Tenon, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Rouen, Rouen
  - CH Alpes Léman, Sallanches
  - CHU Strasbourg, Strasbourg
  - Hopital FOCH, Suresnes
  - CHU toulouse, Toulouse

REFERENCES:
- [Derived] Fakhouri F, Fila M, Hummel A, Ribes D, Sellier-Leclerc AL, Ville S, Pouteil-Noble C, Coindre JP, Le Quintrec M, Rondeau E, Boyer O, Provot F, Djeddi D, Hanf W, Delmas Y, Louillet F, Lahoche A, Favre G, Chatelet V, Launay EA, Presne C, Zaloszyc A, Caillard S, Bally S, Raimbourg Q, Tricot L, Mousson C, Le Thuaut A, Loirat C, Fremeaux-Bacchi V. Eculizumab discontinuation in children and adults with atypical hemolytic-uremic syndrome: a prospective multicenter study. Blood. 2021 May 6;137(18):2438-2449. doi: 10.1182/blood.2020009280. PMID 33270832